CLINICAL TRIAL: NCT00978926
Title: A Study of the Pharmacodynamic Effects of Anti-vascular Endothelial Growth Factor Therapy in Patients With Advanced Malignancies
Status: Completed | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Ross Andrew Soo, National University Hospital, Singapore
Other Study IDs: MC02/15/07
Record Dates: First submitted 2008-06-19; First posted 2009-09-17 (Estimated); Last update posted 2010-04-09 (Estimated); Status verified 2010-04

CONDITIONS: Advanced Malignancy
Keywords: Anti-Vascular Endothelial growth factor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The well-established role of vascular endothelial growth factor (VEGF) in carcinogenesis and tumor angiogenesis has led to the development of agents that target this pathway. Anti-VEGF agents the VEGF monoclonal antibody bevacizumab, and the small molecule VEGF receptor tyrosine kinase inhibitors. Angiogenic factors play a key role in the maintenance of lung integrity and normal endothelial function. Endothelial dysfunction has been implicated in hypertension, proteinuria and retinopathy. One of the major issues of anti-VEGF agents is its long-term toxicity especially taking into account the lack of adequate knowledge in this area and the possibility of prolonged periods of therapy in non-progressing patients. Hypertension and proteinuria are commonly seen in patients treated with anti-VEGF agents. In addition, the investigators have also observed in a relatively high frequency of pulmonary air-filled lesions in patients with malignancy in the lung treated with an anti-VEGF agent. Objectives of this exploratory study are to 1) determine the effect of anti-vascular endothelial growth factor (VEGF) on endothelial function 2) determine endothelial dysfunction as a marker of early response and as an indicator for the development of hypertension and proteinuria 3) characterize the effect of anti-VEGF therapy on the pulmonary function of patients with malignancy (primary or secondary) involving the lung in patients treated with anti-VEGF agents. Pharmacodynamic endpoints to be assessed are: blood pressure, brachial artery reactivity, retinal microvessels, microalbuminuria and proteinuria, pulmonary function, assess the effects of anti-VEGF therapy by assessing brachial artery reactivity, retinal vasculature and pulmonary function in a subset of patients receiving anti-VEGF therapy. The development of markers of endothelial dysfunction may result in the early identification of patients who are non-responders or develop toxicity from anti-VEGF treatment.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility
* Patients who are receiving single agent anti-VEGF therapy
* Signed written informed consent
* Patients with measurable pulmonary malignancy (primary or metastatic) as determined by RECIST will undergo assessment of pulmonary function
* Patients with a known allergy to intravenous contrast used in fluorescein and indocyanine green angiography will be exempt from these investigations but will undergo other study assessments

Exclusion Criteria:

* None

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study aims to assess the pharmacodynamic effects of anti-VEGF therapy. The following groups of patients will be approached:
  Those who are starting on anti-VEGF therapy (such as but not limited to bevacizumab, sunitinib, and sorafenib) as part of routine clinical management or on clinical studies
Sampling Method: Probability Sample
Dates: Start 2009-09

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Ferrara N, Gerber HP, LeCouter J. The biology of VEGF and its receptors. Nat Med. 2003 Jun;9(6):669-76. doi: 10.1038/nm0603-669. PMID 12778165
- [Background] Hicklin DJ, Ellis LM. Role of the vascular endothelial growth factor pathway in tumor growth and angiogenesis. J Clin Oncol. 2005 Feb 10;23(5):1011-27. doi: 10.1200/JCO.2005.06.081. Epub 2004 Dec 7. PMID 15585754